CLINICAL TRIAL: NCT05366556
Title: The Effect of Virtual Reality on Pain and Anxiety During Blood Collection in Adult Patients: Randomized Controlled Trial
Brief Title: The Effect of Virtual Reality on Pain and Anxiety During Blood Collection in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Serap Sayar, Assistant Professor, PhD, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022/009
Record Dates: First submitted 2022-04-29; First posted 2022-05-09 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Adult; Virtual Reality; Anxiety; Pain
Keywords: Adults; Virtual Reality; Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: The adult patients will be divided into two as the experimental and control group. Patients in the experimental group will be informed about the using virtual reality glasses during the taking blood. During this process, their anxiety and pain will be assesed. Patients in the study group will be evaluated 2 times, before the intervention and after the intervention, through data collection tools.
Who Masked: Participant
Masking Description: Single Blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients in the experimental group will be informed about the using virtual reality glasses during the taking blood. During this process, their anxiety and pain will be assesed. Patients in the study group will be evaluated 2 times, before the intervention and after the intervention, through data collection tools.
  Interventions: Behavioral: Virtual reality
- Control group (No Intervention): The control group will receive standard procedure without any intervention

INTERVENTIONS:
Behavioral: Virtual reality — The patient, whose blood will be drawn, will be asked to wear virtual reality glasses after sitting in the blood collection chair. One minute before the start of the blood collection process, "Nature Hiking" will be watched from the virtual reality. Meanwhile, the researcher will complete the preparations for blood collection and will start the blood collection process. It is thought that the blood collection process takes 2-3 minutes on average. During this period, virtual reality will be applied. While blood is being drawn from the patient, the researcher will assess the patient's level of pain with the VAS during the procedure. After the blood draw is completed, the virtual reality glasses will be removed. Then, the patient will be taken to the waiting area and the state anxiety scale will be applied.
  Arms: Experimental group

SUMMARY:
In hospitals, venous blood sampling as the first step in diagnosis and planning of medical treatment is among the most basic and common procedures all over the world. Before the diagnosis and treatment of acute or chronic health problems, venous blood is requested from the doctors and the blood sample is collected by the nurses. Patients experience anxiety for reasons such as the fear of experiencing pain during the blood donation process, fear of seeing blood, and fear that blood-borne diseases will pass. Studies in the literature have generally evaluated the effects on pain and fear by using virtual reality with different techniques in pediatric patients during blood collection, and the relevant research has been reached in adult patients. The aim of this research is to determine the effect of virtual reality on pain and anxiety during blood collection of patients who applied to the blood collection unit of a university hospital.

DETAILED DESCRIPTION:
In hospitals, venous blood sampling as the first step in diagnosis and planning of medical treatment is among the most basic and common procedures all over the world. Before the diagnosis and treatment of acute or chronic health problems, venous blood is requested from the doctors and the blood sample is collected by the nurses. Patients experience anxiety for reasons such as the fear of experiencing pain during the blood donation process, fear of seeing blood and fear that blood-borne diseases will pass. Pain and anxiety because of invasive procedures lead to prolongation of the examination period and treatment procedures, and the rejection of treatment. Various distraction methods such as pharmacological local anesthetic creams, non-pharmacologically vibrating tourniquet, buzzy device, virtual reality have been used to reduce pain during invasive procedures. Vibrating tourniquet application during blood collection in pediatric patients was found to be effective on the pain felt. In another study conducted in pediatric patients, it was found that using a buzzy device, watching cartoons, and playing digital games during blood collection were effective in pain and fear management. Virtual reality is defined as "a technology that allows three-dimensional pictures and animations created in the computer environment to interact with these objects in the environment, which gives the feeling of being in a real environment in people's minds with technological tools". In the studies, virtual reality was applied in many studies during blood collection in pediatric patients. It was found that children who used virtual reality during invasive procedures in the pediatric nephrology clinic reported lower pain intensity and stress level compared to the control group. In the literature, research involving an attempt to reduce pain and anxiety during blood collection in adult patients has been found and studies involving attempts to reduce pain and anxiety during other invasive procedures are limited. In a study examining the pain and fear of adult outpatients during the treatment, it was found that the pain and anxiety levels of the virtual reality application group were low and they were highly satisfied with virtual reality. The aim of this research is to determine the effect of virtual reality on pain and anxiety during blood collection of patients who applied to the blood collection unit of a university hospital.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreed to participate in the research.
* Being 18 years or older
* Being able to read and write Turkish
* No vision and hearing problems
* Not using glasses
* Absence of any psychiatric, cognitive or neurological disease

Exclusion Criteria:

* Patients with visual or hearing impairment
* Patients whose blood cannot be drawn in once

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
State Anxiety Scale mean score | 10 minute
  State Anxiety Scale mean scores of adult patients in the intervention and control groups will be compared before and after the intervention. A minimum of 20 and a maximum of 80 points can be obtained from the scale. If the scale score approaches 80, it indicates high anxiety.
Visual Analog Scale mean score | 2 minute (during the process)
  Mean Visual Analog Scale scores for adult patients of the intervention and control groups will be compared at the time of intervention.The minimum score to be taken from the scale is zero, the maximum score is 10. It shows that the severity of pain increases as the Visual Analog Scale score approaches 10 during blood collection.

CONTACTS AND LOCATIONS:
Overall Officials: Serap SAYAR, PhD, Study Director — KTO Karatay University; Magbul Ahmet Çoban, MScN student, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University Medical Faculty Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The researcher at Necmettin Erbakan University will collect the data